CLINICAL TRIAL: NCT03155633
Title: "Corre, Recupera, Repite, Siempre Saludable".
Brief Title: Run, Recovery, Repeat, Always Healthy ("Corre, Recupera, Repite, Siempre Saludable")
Acronym: CRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: Fundación Trinidad Alfonso (Unknown); Fundación Hospitales NISA (Unknown); SD. Correcaminos (Unknown)
Responsible Party: Principal Investigator, Carlos Hernando, Ph D. Director of Sports Service, Universitat Jaume I
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UJI_CRS001
Record Dates: First submitted 2017-04-26; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Physical Exertion
Keywords: Marathon, runners, biomarkers, recovery

STUDY DESIGN:
Intervention Model Description: The first one performed rests during the 9 days after the race, the second performed continuous race monitored every 48h from the end of the race, and the third group performed aerobic work on an elliptical machine under the same conditions as the group of Continuous race
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rest Group (No Intervention): Rest during the 9 days after the race
- Running Group (Experimental): Running at 95-105% aerobic Threshold on athletics track 48h, 96h, 144h after the race. Control heart devices
  Interventions: Other: Athletics track
- Elliptical Group (Experimental): Running at 95-105% aerobic Threshold on elliptical machine 48h, 96h, 144h after the race. Control heart devices
  Interventions: Other: Elliptical machine

INTERVENTIONS:
Other: Athletics track — Running at 95-105% aerobic Threshold on athletics track 48h, 96h, 144h after the race. Control heart devices
  Arms: Running Group
Other: Elliptical machine — Running at 95-105% aerobic Threshold on elliptical machine 48h, 96h, 144h after the race. Control heart devices
  Arms: Elliptical Group

SUMMARY:
This study has as main objective to know how the processes of recovery are realized after a race of marathon. For this, the participants of a marathon race are divided into three work groups during the 9 days post-marathon, one with rest in the recovery period, another with continuous race three sessions every 48h and another with three sessions of elliptical every 48h .

DETAILED DESCRIPTION:
The marathon runners suffer a high fatigue, as has been studied by different investigations, the proposal of this study is to know how the recovery processes are produced in runners who have completed a 42km test.

To do this, baseline measurements of the runners have been made through stress tests and determinations of biomarkers in blood and urine. Subsequently blood and urine samples were taken the day before the marathon test and blood and urine samples were then taken again on arrival at 24h, 48h, 96h, 144h, and 196h.

At the same time, an intervention was carried out in the recovery phase, with the runners in three groups. The first one performed rests during the 9 days after the race, the second performed continuous race monitored every 48h from the end of the race, and the third group performed aerobic work on an elliptical machine under the same conditions as the group of Continuous race

ELIGIBILITY:
Inclusion Criteria:

* Adults healthy with 30-45 years
* BMI between 16-24,99
* Time in marathon between 3h-4h in men
* Time in marathon between 3h:30min-4h:40min in women

Exclusion Criteria:

* Having heart disease
* Having kidney disease
* Taking a medication on an ongoing basis

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-10-20 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Change in the Blood Physiological parameters | baseline, 0, 24, 48, 96, 144 and 192 hours post-race
  Blood test
Analysis of tne changes in the Physical activity data | One month before the pre-race, accelerometers were worn during seven days. Accelerometers were also worn during nine days starting from the night before the marathon race
  Physical activity measured by wearing accelerometer devices. Physical activity defined as sedentary, light, moderate and vigorous. The aim to wear accelerometers devices is to monitor individuals during recovery time post-marathon race
Change in the Urin Physiological parameters | baseline, 0, 48, 96, 144 and 192 hours post-race
  Urin test

SECONDARY OUTCOMES:
Self-reported questionnaire | One month before the race day
  Personal questionnaire asking for social and training habits
Strength level | pre-marathon race and 0, 48, 96, 144 hours post-marathon race
  Squat Jump (cm). Two jumps per person
Analysis of the change of body mass index | one month before the marathon race day, 24 hours before the marathon race, 2 hours before the marathon race and 10 minutes after the marathon race
  BMI
Physical Condition | One month before the marathon race day
  Maximal oxygen consumption
Body composition | One month before the marathon race day
  Bioimpedance analysis
Heart rate | Through marathon completion, an average of 4 hours
  Recording the number of contractions of the heart per minute (bpm) by using a heart rate monitor during all the marathon race

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Hernando, Principal Investigator — Universitat Jaume I

IPD SHARING:
Plan to Share IPD: Yes
The data are administered by the Investigator Principal, other researchers must request the data they need by written request

REFERENCES:
- [Background] Knechtle B, Nikolaidis PT, Zingg MA, Rosemann T, Rust CA. Differences in age of peak marathon performance between mountain and city marathon running - The 'Jungfrau Marathon' in Switzerland. Chin J Physiol. 2017 Feb 28;60(1):11-22. doi: 10.4077/CJP.2017.BAE400. PMID 28052642
- [Background] Roca E, Nescolarde L, Lupon J, Barallat J, Januzzi JL, Liu P, Cruz Pastor M, Bayes-Genis A. The Dynamics of Cardiovascular Biomarkers in non-Elite Marathon Runners. J Cardiovasc Transl Res. 2017 Apr;10(2):206-208. doi: 10.1007/s12265-017-9744-2. Epub 2017 Apr 5. PMID 28382580
- [Background] Santos VC, Sierra AP, Oliveira R, Cacula KG, Momesso CM, Sato FT, Silva MB, Oliveira HH, Passos ME, de Souza DR, Gondim OS, Benetti M, Levada-Pires AC, Ghorayeb N, Kiss MA, Gorjao R, Pithon-Curi TC, Cury-Boaventura MF. Marathon Race Affects Neutrophil Surface Molecules: Role of Inflammatory Mediators. PLoS One. 2016 Dec 2;11(12):e0166687. doi: 10.1371/journal.pone.0166687. eCollection 2016. PMID 27911915
- [Background] Niemela M, Kangastupa P, Niemela O, Bloigu R, Juvonen T. Individual responses in biomarkers of health after marathon and half-marathon running: is age a factor in troponin changes? Scand J Clin Lab Invest. 2016 Nov;76(7):575-580. doi: 10.1080/00365513.2016.1225122. Epub 2016 Sep 9. PMID 27609306
- [Background] Kim YJ, Ahn JK, Shin KA, Kim CH, Lee YH, Park KM. Correlation of Cardiac Markers and Biomarkers With Blood Pressure of Middle-Aged Marathon Runners. J Clin Hypertens (Greenwich). 2015 Nov;17(11):868-73. doi: 10.1111/jch.12591. Epub 2015 Jun 13. PMID 26073606
- [Background] Tojima M, Noma K, Torii S. Changes in serum creatine kinase, leg muscle tightness, and delayed onset muscle soreness after a full marathon race. J Sports Med Phys Fitness. 2016 Jun;56(6):782-8. Epub 2015 Feb 10. PMID 25665742
- [Background] Knechtle B, Knechtle P, Rosemann T, Lepers R. Personal best marathon time and longest training run, not anthropometry, predict performance in recreational 24-hour ultrarunners. J Strength Cond Res. 2011 Aug;25(8):2212-8. doi: 10.1519/JSC.0b013e3181f6b0c7. PMID 21642857
- [Background] Knechtle B, Knechtle P, Barandun U, Rosemann T, Lepers R. Predictor variables for half marathon race time in recreational female runners. Clinics (Sao Paulo). 2011;66(2):287-91. doi: 10.1590/s1807-59322011000200018. PMID 21484048
- [Derived] Martinez-Navarro I, Montoya-Vieco A, Collado E, Hernando B, Panizo N, Hernando C. Muscle Cramping in the Marathon: Dehydration and Electrolyte Depletion vs. Muscle Damage. J Strength Cond Res. 2022 Jun 1;36(6):1629-1635. doi: 10.1519/JSC.0000000000003713. Epub 2020 Aug 12. PMID 32796418